CLINICAL TRIAL: NCT03282058
Title: The Effect of Silastic Stenting on Post-Operative Intra-Nasal Re-Mucosalization
Brief Title: Silastic Stent Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Arif Janjua, MD, FRCSC, Otolarynology - Head & Neck Surgery; Endoscopic Sinus & Skull Based Surgery, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H14-02101
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Pituitary Tumour
Keywords: Silastic Stenting; Trans-nasal Endoscopic Surgery; Post-operative Intra-nasal Re-mucosalization
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in one of two groups (stent vs no stent).
Who Masked: Outcomes Assessor
Masking Description: Histology of the healing tissues will be examined by a pathologist who is blinded to whether the patient received or did not receive stenting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silastic Stent (Experimental): At the time of surgery, if the patient is identified in the "silastic stent" arm, dressing of the septal donor site with silastic stents will be performed after reconstruction has been achieved and the surgeon feels that the surgery proceeded routinely.
  Interventions: Device: Silastic Stent
- No Stent (No Intervention): At the time of surgery, if the patient is identified in the "no silastic stent" arm, dressing of the septal donor site without the stent will be performed after reconstruction has been achieved and the surgeon feels that the surgery proceeded routinely - this is currently the standard of care.

INTERVENTIONS:
Device: Silastic Stent — The silastic stent is a splint made of silicone.
  Arms: Silastic Stent

SUMMARY:
Endoscopic skull base surgery is a relatively new procedure that is now a standard of care for surgeries at the base of the skull; however there are no studies that examine the healing process of the nasal lining with the use of silastic (silicone) stents (or splints) that might be placed at the time of surgery. While there is some evidence to suggest that the use of stents improves wound healing, the decision to use a stent or not is currently up to the preference of the surgeon. To investigate the impact of stents on post-surgical healing, the investigators at Vancouver General Hospital will compare patients undergoing trans-sphenoidal pituitary surgeries with septal flap reconstruction with the use of silastic stents to line the septal donor site, and compare their recovery to those who did not receive stents. The investigators hypothesize that the use of silastic stents in endonasal surgery increases the rate of mucosal healing, and better quality mucosal regeneration, and with no effect on the patients experience after surgery. In this randomized control trial the investigators aim to recruit 26 (13 in each arm) study participants. The primary outcome is to determine the effect of silastic stunting on healing of the naso-septal flap donor site. This objective will be achieved by assessment of endoscopic photographs of healing tissue and histologic assessment of healing tissues. The secondary outcome involves questionnaires that measure the patient's subjective nasal symptoms prior to and following endoscopic skull based surgery. Total time commitment for the study participant is about 4 months across 4 study visits (all of which are part of standard of care): the assessment visit, surgery, 4 weeks post-operative follow up visit and 12 week post-operative follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing trans-sphenoidal endoscopic pituitary surgery at their first post-operative appointment

Exclusion Criteria:

* patients with inflammatory sinus conditions
* patients having undergone extensive skull base reconstructions
* patients having received previous radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-04-04 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining the effect of silastic stunting on gross level healing of the naso-septal flap donor sites in two aspects gross level healing and microscopic level of healing. | Total time approx. 4 months (pre-operative assessment; surgery; 4 and 12 weeks post-operative follow up appointments)
  Visual assessment of endoscopic photographs of healing tissue.
Determining the effect of silastic stunting on microscopic level healing of the naso-septal flap donor sites in two aspects gross level healing and microscopic level of healing. | Total time approx. 4 months (pre-operative assessment; surgery; 4 and 12 weeks post-operative follow up appointments)
  Histologic assessment of healing tissues.
Determining the effect of silastic stunting on nasa-septal flap donor sites on the patient's subjective nasal symptoms following endoscopic skull based surgery. | Total time approx. 4 months (pre-operative assessment; surgery; 4 and 12 weeks post-operative follow up appointments)
  Participants will fill out a quality of life questionnaire called Sino-Nasal Outcome Test (SNOT-22).
Determining the effect of silastic stunting on nasa-septal flap donor sites on the patient's subjective post-operative outcomes following endoscopic skull based surgery. | Total time approx. 4 months (post-operative follow up at 4 and 12 weeks)
  Participants will fill out a post-operative rating scale.
Physician's evaluation of the effect of silastic stunting on nasa-septal flap donor sites following endoscopic skull based surgery. | Total time approx. 4 months (surgery; post-operative follow up at 4 and 12 weeks)
  Physician will fill out an outcome measures evaluation scale.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Janjua, MD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bednarski KA, Kuhn FA. Stents and drug-eluting stents. Otolaryngol Clin North Am. 2009 Oct;42(5):857-66, x. doi: 10.1016/j.otc.2009.07.001. PMID 19909864
- [Background] Cowin A, McIntosh D, Wormald PJ. Healing of wounds created in the nasal mucosa following endoscopic sinus surgery can be affected by different nasal packing materials. Primary Intention Vol. 10 No. 3 August 2002.
- [Background] Gamoletti R, Lanzarini P, Sanna M, Zini C. Regenerated middle ear mucosa after tympanoplasty. Part II. Scanning electron microscopy. Otolaryngol Head Neck Surg. 1986 Apr;94(4):430-4. doi: 10.1177/019459988609400404. PMID 3086802
- [Background] Ng M, Linthicum FH Jr. Long-term effects of Silastic sheeting in the middle ear. Laryngoscope. 1992 Oct;102(10):1097-102. doi: 10.1288/00005537-199210000-00002. PMID 1328786
- [Background] Soper, D.S. (2014). A-priori Sample Size Calculator for Student t-Tests [Software]. Available from http://www.danielsoper.com/statcalc